CLINICAL TRIAL: NCT04503096
Title: High-dose Accelerated Repetitive Transcranial Magnetic Stimulation to Cognitive Control Neurocircuitry in Mild Cognitive Impairment: A Safety and Feasibility Study
Brief Title: Plasticity Using Stimulation and Habit: A Pilot Open-label rTMS Study for MCI
Acronym: PUSH-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center of Neuromodulation for Rehabilitation (Other)
Responsible Party: Principal Investigator, Andreana Benitez, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100536
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- High-dose accelerated rTMS (Experimental)
  Interventions: Device: High-dose accelerated rTMS

INTERVENTIONS:
Device: High-dose accelerated rTMS — A MagVenture MagPro Transcranial Magnetic Stimulation (TMS) System will be utilized. All participants will receive open-label treatment for approximately eight, 3-minute sessions of intermittent theta burst rTMS on each of three days within an eight-day span. A single session = 600 pulses at 120% resting motor threshold (rMT), intermittent Theta Burst Stimulation (iTBS) triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 s to left dorsolateral prefrontal cortex. Total pulses = 14,400. To enable adherence and retention, the days do not need to be contiguous. Same day sessions will be separated by 10-15 minutes, but more accounting for participant comfort.

SUMMARY:
The goal of this pilot study is to determine whether a high-dose form of non-invasive brain stimulation is a promising and safe treatment for Mild Cognitive Impairment (MCI). Transcranial magnetic stimulation (TMS) is an FDA approved treatment for depression. In studies of TMS for depression and other disorders, individuals have experienced improved cognitive function. Thus, the current study is testing whether TMS is safe, feasible and effective in improving cognition in individuals with MCI.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-85
* English as a first/primary language
* Has been diagnosed with MCI by a healthcare provider within the past two years per National Institute on Aging - Alzheimer's Association (NIA-AA) criteria: (1) Concern regarding cognitive decline reported by patient, informant, or clinician, (2) Objective evidence of impairment for age in 1+ cognitive domains, typically memory, (3) Preserved independent function, (4) no dementia.
* Has met actuarial neuropsychological criteria for amnestic MCI: (1) ≥2 impaired scores (i.e. ≤16th %ile) within one cognitive domain, or (2) ≥1 impaired scores (i.e. ≤16th %ile) in ≥3 cognitive domains, using demographically-corrected normative data. (1) and (2) must include the Memory domain.
* The primary suspected etiology of amnestic MCI must be neurodegenerative, with competing differential diagnoses (e.g. psychiatric disorder, movement disorder, reversible causes, substance use) ruled out as the primary etiology/ies following a clinical evaluation by a healthcare provider.
* Ability to provide independent informed consent, consistent with the MCI diagnostic criterion of preserved independent function.

Exclusion Criteria:

* Dementia diagnosis per the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) or NIA-AA criteria.
* Daily/weekly use of anticholinergics, neuroleptics, sedatives, or bupropion. Stimulant use may be allowed pending investigator review. Cholinesterase inhibitors, NMDA receptor antagonists, and antidepressants are allowed if on a stable regimen of four weeks prior to enrollment.
* History of significant or unstable condition/s that may impact cognition such as significant cardiac, cerebrovascular, or metabolic disease, severe mental illness (e.g. bipolar disorder, psychoses), alcohol or substance use disorder, developmental disorder, or other neurologic disease (e.g. severe brain injury, seizures).
* MRI and TMS contraindications (e.g., implants, claustrophobia, conditions/treatments that lower seizure threshold, taking medications that have short half-lives, no quantifiable motor threshold, active substance use disorder, bipolar disorder).
* Is enrolled in a clinical trial and/or has received an investigational medication within the last 30 days.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreana Benitez, PhD, Principal Investigator — Medical University of South Carolina; Lisa McTeague, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aghamoosa S, Lopez J, Rbeiz K, Fleischmann HH, Horn O, Madden K, Caulfield KA, Antonucci MU, Revuelta G, McTeague LM, Benitez A. A phase I trial of accelerated intermittent theta burst rTMS for amnestic MCI. J Neurol Neurosurg Psychiatry. 2024 Oct 16;95(11):1036-1045. doi: 10.1136/jnnp-2023-332680. PMID 38719432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were referred by neurologists and neuropsychologists at MUSC's outpatient memory disorders and neuropsychology clinics. They were recruited between 12/22/2020 and 5/5/2022. The first participant was enrolled on 4/12/2021 and the last participant was enrolled on 6/1/2022.
Pre-assignment Details: Of the 67 participants assessed for eligibility, 10 did not meet inclusion criteria, 15 met exclusion criteria, 17 declined to participate, and 1 was excluded for other reasons. 24 participants were assigned to treatment.
Groups:
- High-dose Accelerated rTMS: High-dose accelerated rTMS: A MagVenture MagPro Transcranial Magnetic Stimulation (TMS) System will be utilized. All participants will receive open-label treatment for approximately eight, 3-minute sessions of intermittent theta burst rTMS on each of three days within an eight-day span. A single session = 600 pulses at 120% rMT, intermittent Theta Burst Stimulation (iTBS) triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 s to left dorsolateral prefrontal cortex. Total pulses = 14,400. To enable adherence and retention, the days do not need to be contiguous. Same day sessions will be separated by 10-15 minutes, but more accounting for participant comfort.
Period: Overall Study
Arm/Group | High-dose Accelerated rTMS
Started | 24
Completed | 21
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | High-dose Accelerated rTMS
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: Z-score] — The MoCA is a psychometrist-administered brief cognitive assessment tool with raw total scores ranging from 0 to 30, with higher values indicating better cognition. For this analysis raw total scores were converted to age- and education-adjusted Z-scores using published norms (Rossetti et al., 2011). Z-scores have a mean of 0 and a standard deviation of 1. Lower scores indicate worse performance. Population: This includes only participants with both pre- and post-treatment data.
  Z-score
    number analyzed (Participants) | 21
    (all) | -1.25 (1.38)
Hamilton Depression Rating Scale (HAM-D) [Mean (Standard Deviation); unit: scores on a scale] — The Hamilton Depression Rating Scale (Ham-D) is a 17-item interviewer-administered structured questionnaire designed to assess symptoms of depression with scores ranging from 0 to 53, with higher scores indicating more depressive symptoms. Population: This includes only participants with both pre- and post-treatment data.
  scores on a scale
    number analyzed (Participants) | 21
    (all) | .24 (.77)
Geriatric Depression Scale (GDS) [Mean (Standard Deviation); unit: scores on a scale] — The Geriatric Depression Scale (GDS) is a 30-item scale that evaluates the severity of depressive symptoms in older adults with scores ranging from 0 to 30, with higher scores indicating more depressive symptoms. Population: This includes only participants with both pre- and post-treatment data.
  scores on a scale
    number analyzed (Participants) | 20
    (all) | 4.55 (3.14)
Fluid Cognition Composite [Mean (Standard Deviation); unit: T-score] — Fluid cognition was measured using the iPad-administered NIH Toolbox Cognition Battery (NIHTB-CB). Fluid Cognition Composite scores were calculated by averaging the demographically adjusted (age, education, sex, race/ethnicity; Casaletto et al., 2015) T-scores for 4 NIHTB-CB tests: flanker inhibitory control, list sorting working memory, pattern comparison processing speed, and dimensional change card sort. T-Scores have a mean of 50 and a standard deviation of 10. Lower scores indicate worse performance. Population: This includes only participants with both pre- and post-treatment data.
  T-score
    number analyzed (Participants) | 21
    (all) | 40.25 (8.07)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Structural Brain Change on T1- and T2-weighted Magnetic Resonance Imaging (MRI)
Description: Clinically significant structural brain change were determined by a board-certified neuroradiologist who reviewed both the pre-treatment and post-treatment structural (T1- and T2-weighted) MRI scans to identify the presence of any changes from pre- to post-treatment based on their clinical read of the images.
Time Frame: Baseline prior to treatment and at follow-up within 1 week post-treatment
Population: Participants who completed both the pre- and post-treatment assessments were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Accelerated rTMS
Number analyzed (Participants) | 21
Participants | 0

2. Primary Outcome: Change From Baseline Global Cognition, as Measured by the Montreal Cognitive Assessment (MoCA)
Description: The MoCA is a psychometrist-administered brief cognitive assessment tool with raw total scores ranging from 0 to 30, with higher values indicating better cognition. For this analysis raw total scores were converted to age- and education-adjusted Z-scores using published norms (Rossetti et al., 2011). Z-scores have a mean of 0 and a standard deviation of 1. Lower scores indicate worse performance. The outcome measure reported below is the mean Z-score score at the 1-week post-treatment assessment. The statistical analysis compares this mean score to the mean score at Baseline.
Time Frame: Baseline prior to treatment and at follow-up within 1 week post-treatment
Population: Participants who completed both the pre- and post-treatment assessments were included in this analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | High-dose Accelerated rTMS
Number analyzed (Participants) | 21
Z-score | -1.20 (1.18)
Statistical Analysis 1: Comparison: High-dose Accelerated rTMS; Test type: Other — To monitor safety, paired t-tests were conducted to test for pre- to post-treatment differences in global cognition (i.e., MoCA z-scores); p = 0.725, t-test, 2 sided

3. Primary Outcome: Change in the Review of Systems Criteria Compared to Baseline
Description: A review of systems questionnaire will be administered to rate the subjective symptom (headache, scalp pain, arm/hand pain, other pain(s), numbness/tingling, other sensation(s), weakness, loss of dexterity, vision/hearing change(s), ear ringing, nausea/vomiting, appetite loss, rash, skin change(s) or any other symptom(s)) on a scale of 0 to 5 (none, minimal, mild, moderate, marked, severe).
Time Frame: Baseline prior to treatment and at follow-up within 1 week post-treatment
Population: Participants who completed both the pre- and post-treatment assessments were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Accelerated rTMS
Number analyzed (Participants) | 21
Participants
  Headache: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Headache: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Headache: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Headache: Post-Treatment: Minimal/none (0-1) | 20
  Headache: Post-Treatment: Mild/moderate (2-3) | 1
  Headache: Post-Treatment: Marked/severe (4-5) | 0
  Scalp pain: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Scalp pain: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Scalp pain: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Scalp pain: Post-Treatment: Minimal/none (0-1) | 19
  Scalp pain: Post-Treatment: Mild/moderate (2-3) | 2
  Scalp pain: Post-Treatment: Marked/severe (4-5) | 0
  Arm/hand pain: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Arm/hand pain: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Arm/hand pain: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Arm/hand pain: Post-Treatment: Minimal/none (0-1) | 21
  Arm/hand pain: Post-Treatment: Mild/moderate (2-3) | 0
  Arm/hand pain: Post-Treatment: Marked/severe (4-5) | 0
  Other pain: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Other pain: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Other pain: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Other pain: Post-Treatment: Minimal/none (0-1) | 20
  Other pain: Post-Treatment: Mild/moderate (2-3) | 1
  Other pain: Post-Treatment: Marked/severe (4-5) | 0
  Weakness: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Weakness: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Weakness: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Weakness: Post-Treatment: Minimal/none (0-1) | 21
  Weakness: Post-Treatment: Mild/moderate (2-3) | 0
  Weakness: Post-Treatment: Marked/severe (4-5) | 0
  Loss of dexterity: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Loss of dexterity: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Loss of dexterity: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Loss of dexterity: Post-Treatment: Minimal/none (0-1) | 21
  Loss of dexterity: Post-Treatment: Mild/moderate (2-3) | 0
  Loss of dexterity: Post-Treatment: Marked/severe (4-5) | 0
  Vision changes: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Vision changes: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Vision changes: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Vision changes: Post-Treatment: Minimal/none (0-1) | 21
  Vision changes: Post-Treatment: Mild/moderate (2-3) | 0
  Vision changes: Post-Treatment: Marked/severe (4-5) | 0
  Hearing changes: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Hearing changes: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Hearing changes: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Hearing changes: Post-Treatment: Minimal/none (0-1) | 19
  Hearing changes: Post-Treatment: Mild/moderate (2-3) | 2
  Hearing changes: Post-Treatment: Marked/severe (4-5) | 0
  Ear ringing: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Ear ringing: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Ear ringing: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Ear ringing: Post-Treatment: Minimal/none (0-1) | 20
  Ear ringing: Post-Treatment: Mild/moderate (2-3) | 1
  Ear ringing: Post-Treatment: Marked/severe (4-5) | 0
  Nausea/Vomiting: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Nausea/Vomiting: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Nausea/Vomiting: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Nausea/Vomiting: Post-Treatment: Minimal/none (0-1) | 21
  Nausea/Vomiting: Post-Treatment: Mild/moderate (2-3) | 0
  Nausea/Vomiting: Post-Treatment: Marked/severe (4-5) | 0
  Appetite loss: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Appetite loss: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Appetite loss: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Appetite loss: Post-Treatment: Minimal/none (0-1) | 21
  Appetite loss: Post-Treatment: Mild/moderate (2-3) | 0
  Appetite loss: Post-Treatment: Marked/severe (4-5) | 0
  Rash: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Rash: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Rash: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Rash: Post-Treatment: Minimal/none (0-1) | 21
  Rash: Post-Treatment: Mild/moderate (2-3) | 0
  Rash: Post-Treatment: Marked/severe (4-5) | 0
  Skin changes: Treatment day 1 (Baseline): Minimal/none (0-1) | 21
  Skin changes: Treatment day 1 (Baseline): Mild/moderate (2-3) | 0
  Skin changes: Treatment day 1 (Baseline): Marked/severe (4-5) | 0
  Skin changes: Post-Treatment: Minimal/none (0-1) | 21
  Skin changes: Post-Treatment: Mild/moderate (2-3) | 0
  Skin changes: Post-Treatment: Marked/severe (4-5) | 0

4. Primary Outcome: Patient Perception of Treatment Acceptability
Description: A 15-item study-specific questionnaire of rTMS treatment acceptability, with each item rated on a scale from 1 to 5 (1 = not at all, 3 = somewhat, 5 = very much so). Higher scores indicate better acceptability for the first 10 items, lower scores indicate better acceptability for the last 5 items.
Time Frame: Administered at post-treatment
Population: Participants who completed both the pre- and post-treatment assessments were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | High-dose Accelerated rTMS
Number analyzed (Participants) | 21
score on a scale
  "I was motivated to attend the rTMS sessions." | 5 [4 to 5]
  "I was committed to completing the treatment course." | 5 [5 to 5]
  "I was interested in the rTMS techniques and learning about them." | 5 [5 to 5]
  "I understand the purpose of the treatment and how it could help my symptoms." | 5 [5 to 5]
  "I would be open to completing another course of rTMS treatment in the future, if needed." | 5 [5 to 5]
  "The rTMS treatment helped improve my ability to cope with daily challenges." | 3 [2 to 4]
  Paraphrased: Condensed treatment was preferable to conventional treatment course | 5 [5 to 5]
  "The staff members were attentive and sensitive to my needs during treatment." | 5 [5 to 5]
  "The staff members explained all procedures to me and answered my questions." | 5 [5 to 5]
  "There was plenty of flexibility in scheduling rTMS sessions around my other obligations." | 5 [5 to 5]
  "At times I wanted to quit treatment." | 1 [1 to 1]
  "Treatment sessions were stressful." | 1 [1 to 2]
  "It was hard to stay awake during the rTMS sessions." | 1 [1 to 1]
  "I experienced pain and discomfort during treatment that was difficult to tolerate." | 1 [1 to 1]
  "Completing multiple rTMS sessions in each day was at times tiring." | 1 [1 to 2]

5. Primary Outcome: Retention Rate
Description: Percentage of participants who completed the study (n=21) relative to all participants who initiated treatment (n=22).
Time Frame: Baseline prior to treatment and at follow-up within 1 week post-treatment
Population: All participants who initiated treatment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Accelerated rTMS
Number analyzed (Participants) | 22
Participants | 21

6. Secondary Outcome: Change From Baseline Depression, as Measured by the Hamilton Depression Rating Scale (HAM-D)
Description: The Hamilton Depression Rating Scale (Ham-D) is a 17-item interviewer-administered structured questionnaire designed to assess symptoms of depression with scores ranging from 0 to 53, with higher scores indicating more depressive symptoms. The outcome measure reported below is the mean score at the 1-week post-treatment assessment. The statistical analysis compares this mean score to the mean score at Baseline.
Time Frame: Baseline prior to treatment and at follow-up within 1 week post-treatment
Population: Participants who completed both the pre- and post-treatment assessments were included in this analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High-dose Accelerated rTMS
Number analyzed (Participants) | 21
scores on a scale | .33 (.91)
Statistical Analysis 1: Comparison: High-dose Accelerated rTMS; Test type: Other — Paired t-tests were conducted to test for pre- to post-treatment changes in depression using HAM-D raw scores; p = .605, t-test, 2 sided

7. Secondary Outcome: Change From Baseline Depression, as Measured by the Geriatric Depression Scale (GDS)
Description: The Geriatric Depression Scale (GDS) is a 30-item scale that evaluates the severity of depressive symptoms in older adults with scores ranging from 0 to 30, with higher scores indicating more depressive symptoms. The outcome measure reported below is the mean score at the 1-week post-treatment assessment. The statistical analysis compares this mean score to the mean score at Baseline.
Time Frame: Baseline prior to treatment and at follow-up within 1 week post-treatment
Population: Participants who completed both the pre- and post-treatment assessments were included in this analysis. Of the 21 participants who completed treatment, one was missing a GDS score.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High-dose Accelerated rTMS
Number analyzed (Participants) | 20
scores on a scale | 4.65 (3.11)
Statistical Analysis 1: Comparison: High-dose Accelerated rTMS; Test type: Other — Paired t-tests were conducted to test for pre- to post-treatment changes in depression using GDS raw scores; p = .897, t-test, 2 sided

8. Secondary Outcome: Change From Baseline Cognition, as Measured by the Fluid Cognition Composite Score From the NIH Toolbox Cognition Battery
Description: Fluid cognition was measured using the iPad-administered NIH Toolbox Cognition Battery (NIHTB-CB). Fluid Cognition Composite scores were calculated by averaging the demographically adjusted (age, education, sex, race/ethnicity; Casaletto et al., 2015) T-scores for 4 NIHTB-CB tests: the flanker inhibitory control, list sorting working memory, pattern comparison processing speed, and dimensional change card sort tests. T-Scores have a mean of 50 and a standard deviation of 10. Lower scores indicate worse performance. The outcome measure reported below is the mean T-score at the 1-week post-treatment assessment. The statistical analysis compares this mean score to the mean score at Baseline.
Time Frame: Baseline prior to treatment and at follow-up within 1 week post-treatment
Population: Participants who completed both the pre- and post-treatment assessments were included in this analysis.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | High-dose Accelerated rTMS
Number analyzed (Participants) | 21
T-score | 43.67 (7.85)
Statistical Analysis 1: Comparison: High-dose Accelerated rTMS; Test type: Other — Paired t-tests were conducted to test for pre- to post-treatment changes in cognition using Fluid Cognition Composite Scores; p < .001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: In this study, other (i.e., non-serious) adverse events were defined as those that were 1) unexpected, 2) related or possibly related to study participation, AND 3) serious or more prevalent than expected. This definition was approved by our local Institutional Review Board (IRB).
Arm/Group | High-dose Accelerated rTMS
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT04503096/Prot_SAP_003.pdf
  • Informed Consent Form (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT04503096/ICF_004.pdf